CLINICAL TRIAL: NCT03089918
Title: An Open-Label Microdosing Study to Investigate the Regional Brain Kinetics of Brain Drug Transporters Using P-glycoprotein and Breast Cancer Resistance Protein Substrates and by Using the Positron Emission Tomography Ligand 11C-JNJ-63779586 in the Human Brain
Brief Title: A Study to Investigate the Regional Brain Kinetics of Brain Drug Transporters Using P-glycoprotein and Breast Cancer Resistance Protein Substrates and by Using the Positron Emission Tomography Ligand 11C-JNJ-63779586 in the Human Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR108288; 63779586NAP1001 (Other: Janssen Research & Development, LLC); 2016-001756-21 (EudraCT Number)
Record Dates: First submitted 2017-03-21; First posted 2017-03-24 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Healthy Adult Male Participants) (Experimental): Participants will receive intravenous (IV) injection with 370 megabecquerel (MBq) 11C-JNJ-63779586 on Day 1 of Part A.
  Interventions: Drug: 11C-JNJ-63779586
- Part B (Mild AD and Healthy age- and Gender-Matched Controls) (Experimental): Participants will receive single IV injection of 11C-JNJ-63779586 on Day 1 of Part B followed by saline flush. During Part B, the dose may be reduced based on whole body dosimetric findings and image quality seen in Part A.
  Interventions: Drug: 11C-JNJ-63779586

INTERVENTIONS:
Drug: 11C-JNJ-63779586 — Participants will receive IV injection with 11C-JNJ-63779586 in Part A and Part B.

SUMMARY:
The purpose of this study is to investigate the total body biodistribution and radiation dosimetry of 11C-JNJ-63779586 by Positron Emission Tomography (PET) in healthy young adult males (Part A); to estimate and compare the uptake, distribution, and clearance of 11C-JNJ-63779586 in the brain by PET between mild Alzheimer Disease (AD) participants (males/females) and age- and gender-matched control participants (Part B), corrected for regional cerebral blood flow differences; and to model the tissue specific kinetics of 11C-JNJ-63779586 in human brain with the appropriate input function (IF) (Part B).

ELIGIBILITY:
Inclusion Criteria:

Part A

* Healthy men between 18 and 55 years of age, inclusive
* Body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2) ², inclusive, and a body weight of not less than 50 kilogram (kg) Part B
* Men or women with mild Alzheimer's Disease (AD), age- and gender-matched control participants, between 55 and 85 years of age, inclusive
* BMI between 18 and 35 kg/m^2, inclusive, and a body weight of not less than 50 kg
* Mild AD participants will be amyloid positive and have a mini-mental state examination (MMSE) greater than or equal to (>=) 20. The matched control participants will be amyloid negative and have a MMSE >= 26, respectively

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency (estimated glomerular filtration rate [eGFR] within the screening period of less than 60 milliLitre per minute per 1.73 meter square [mL/min/1.73 m^2], thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study center as deemed appropriate by the investigator
* Participant has a clinically relevant abnormal physical- or neurological examination, vital signs or 12-lead electrocardiogram (ECG)
* Participant has a history of epilepsy or fits or unexplained black-outs other than vasovagal collapse within 10 years before screening
* Participant has past or planned exposure to ionizing radiation that in combination with the planned administration with the study Positron Emission Tomography (PET) ligand and Computerized Tomography (CT) scan would result in a cumulative exposure that exceeds local recommended exposure limits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Effective Radiation Dose Following Injection of 11C-JNJ-63779586 (Part A) | Day 1
  Whole body and organ specific dosimetry for the tracer will be estimated using specific software for calculation of the absorbed radiation dose. Afterwards, dosimetry will be compared with other carbon-11 labeled radiotracers. According to these results, the same or lower dose might be used for Part B, to prevent high radiation doses to certain organs.
Total and Regional Brain Compartmental Kinetics for Volume of Distribution of 11C-JNJ-63779586 (Part B) | Day 1
  Regional brain uptake will be determined using a Volume of interest (VOI) based analysis. Differences in regional brain uptake between Alzheimer Disease (AD) and control participants will be determined using statistical parametric mapping. Regional uptake of 11C-JNJ-63779586 into brain (K1) will be assessed and compared between participants with AD and control participants, corrected for regional blood flow.
Percent Intact Tracer of 11C-JNJ-63779586 in Blood Samples (Part B) | Day 1
  Sequential arterial blood samples will be taken post tracer injection to model an arterial input function (IF) of the tracer and allow analysis of radio metabolites (percent intact tracer).
Radiometabolite Fraction of 11C-JNJ-63779586 in Blood Samples (Part B) | Day 1
  Sequential arterial blood samples will be taken post tracer injection to model an arterial input function (IF) of the tracer and allow analysis of radio metabolites (percent intact tracer).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability (Part A and Part B) | Up to 29 days (Part A) and Up to 105 days (Part B)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- Belgium (2):
  - UZ Leuven, Leuven
  - University of Antwerpen, Wilrijk